CLINICAL TRIAL: NCT05400447
Title: Multicenter, Prospective, Observational Post Market Clinical Follow-up Study to Evaluate Safety of TIPMED TPM08 Total Knee Prosthesis Systems and TPM Revision Knee Prosthesis Systems
Brief Title: PMCF Study to Evaluate Safety of TIPMED TPM08 Total Knee Prosthesis Systems and TPM Revision Knee Prosthesis Systems
Status: Completed | Type: Observational
Sponsor: TIPMED Medical Device Manufacturing Ltd. Co. (Industry)
Responsible Party: Sponsor
Other Study IDs: INFO TPM08
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Knee Arthroplasty
Keywords: Knee Prosthesis; Total Knee Arthroplasty; Revision Knee Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a observational multicenter study to assess the safety of TIPMED TPM08 Total Knee Prosthesis Systems and TPM Revision Knee Prosthesis Systems used for total knee arthroplasty or revision knee arthroplasty.

DETAILED DESCRIPTION:
In this study, short term (12 months) safety data of TIPMED TPM08 Total Knee Prosthesis System and TPM Revision Knee Prosthesis System will be evaluated using Case Report Forms (CRF). A CRF should be completed at each control visit of the participants by investigator in order to assess safety of the TIPMED Knee Prosthesis Systems by success of operation, occurrence of adverse events during procedure or as the effects in 12 months period resulting from TIPMED Knee Prosthesis Systems. CRF will also include questions related to performance and effectiveness of TIPMED Knee Prosthesis Systems.

Participants should be treated according to instructions-for-use of the implants and accessories and according to clinical routine. The devices must have been used exclusively by physicians who are experienced in knee arthroplasty techniques and who are experienced in using the products in operations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged older than 18 years of age,
* The subjects with appropriate indication for primary total or revision knee arthroplasty,
* The subjects who used TIPMED TPM08 Primary Total or Revision Knee Prosthesis System in their surgery,
* Subjects not under legal disability,
* Subjects or guardian who is willing and able to sign the informed consent form.

Exclusion Criteria:

- Subjects in another interventional clinical trial will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients, who agree to participate in the study, treated with TIPMED TPM08 Primary Total or Revision Knee Prosthesis Systems will be included.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Safety data | 12 months
  Assessment of safety data during 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Salih Kemal Aktuglu, Study Director — Ege University Hospital
Locations (5):
- Turkey (Türkiye) (5):
  - Republic of Turkey Ministry of Health Balıkesir Provincial Health Directorate Ataturk City Hospital, Balıkesir, Altıeylül
  - Ege University Hospital, Izmir, Bornova
  - Republic of Turkey Ministry of Health Izmir Provincial Health Directorate Buca Seyfi Demirsoy Training And Research Hospital, Izmir, Buca
  - Republic of Turkey Ministry of Health Balıkesir Provincial Health Directorate Burhaniye Public Hospital, Balıkesir, Burhaniye
  - Republic of Turkey Ministry of Health Izmir Provincial Health Directorate Menemen Public Hospital, Izmir, Menemen